CLINICAL TRIAL: NCT04835402
Title: A Phase II Study of Electroporation Potentiated Immunotherapy in Liver Metastatic
Brief Title: Electroporation Potentiated Immunotherapy in Cancer
Acronym: EPIC-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Collaborators: Odense University Hospital (Other); Aalborg University (Other); Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor of surgery, Consultant surgeon, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIC-1; 2020-004536-22 (EudraCT Number); N-20200085 (Other: The North Denmark Region Committee on Health Research Ethics)
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Pancreas Cancer, Metastatic
Keywords: Irreversible electroporation; Pembrolizumab; Immune checkpoint inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Day 1: Pembrolizumab 400mg Day 10: Irreversible electroporation Day 42/84/126/168: Pembrolizumab 400mg
  Interventions: Drug: Pembrolizumab; Device: Irreversible electroporation

INTERVENTIONS:
Drug: Pembrolizumab — 400mg every 6 weeks
  Other Names: Irreversible electroporation (NanoKnife(tm), Angiodynamics)
Device: Irreversible electroporation — Percutaneous ablation of one liver metastasis
  Other Names: NanoKnife(tm) (Angiodynamics)

SUMMARY:
The study is investigating the efficacy and safety of combined irreversible electroporation (IRE) and checkpoint inhibition in metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether checkpoint inhibition in conjunction with IRE of a single liver metastasis can elicit a systemic anticancer immune response in patients with pancreatic cancer.

Adult patients, in WHO performance status 0-1, with liver metastatic pancreatic cancer, intolerant to or progressing on first or further lines of chemotherapy can enter the trial. Pembrolizumab infusion is given every six weeks for up to six months. IRE of a single liver metastasis is performed between the first and second pembrolizumab infusion.

Response to the therapy is examined by CT (RECIST) on non-IRE-ablated lesions every 2 months. Assessments of changes in peripheral blood immune cell composition, tumor gene expression and tumor infiltrating lymphocytes is performed on serial biopsies and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified pancreatic adenocarcinoma, based on either a biopsy of the primary tumor or a metastasis
2. One liver metastasis treatable by IRE (as determined by MDT at Aalborg University Hospital)
3. One tumor lesion suited for repeated biopsy by transcutaneous core needle (preferably another lesion than that used for IRE)
4. At least one measurable lesion (RECIST version 1.1) other than the liver metastasis to be treated by IRE
5. At least one course of chemotherapy for metastatic or inoperable disease discontinued due to treatment failure or intolerance
6. Performance status 0-1
7. ASA ≤ 3
8. ≥ 18 years of age
9. Written and orally informed consent
10. Sufficient available histological tumor material stored in biobank or obtainable by new biopsy
11. Patient acceptance of collection of blood samples for translational research and two additional biopsies during treatment
12. Adequate bone marrow function, liver function, and renal function (within 7 days prior to enrollment):

    1. Neutrophils (ANC) ≥ 1.5 x 109/l
    2. Platelet count ≥ 100 x 109/l
    3. Hemoglobin ≥ 6 mmol/l
    4. Plasma bilirubin ≤ 1.5 x ULN
    5. Plasma alanine transaminase (ALAT) < 5 x ULN
    6. Plasma creatinine ≤ 1.5 x ULN
    7. INR ≤ 1.5

Exclusion Criteria:

1. Underlying medical disease not adequately treated (e.g. poorly regulated diabetes and symptomatic cardiac disease)
2. Prior or current autoimmune disorder with risk of serious toxicity during treatment with checkpoint inhibitor
3. Acute myocardial infarction, cerebral vascular attack, transient ischemic attack or subarachnoid hemorrhage within 6 months from start of treatment
4. Previous reception of allogeneic stem cells or solid organ donation
5. Active infection requiring systemic therapy within 7 days prior to treatment initiation
6. Positive HIV, HBV, and HCV test results (prior testing or new testing in patients at risk)
7. Active psychiatric disease or history of drug or alcohol abuse affecting participation
8. Allergy to active substance or any of the auxiliary agents, including known severe allergy to anesthetic agent, paralytic agent or any of the equipment used during treatment
9. Expected need for systemic corticosteroid or other systemic immunosuppressive drug during the course of this clinical trial. A low dose of e.g. prednisone ≤ 10 mg/day is permitted for maximally 7 consecutive days
10. Coexisting malignant disease, except non-melanoma skin cancer
11. Symptomatic or untreated CNS metastases
12. Liver cirrhosis Child Pugh >A
13. Pregnant or breast-feeding patients. For women of childbearing potential, a negative pregnancy test (minimum sensitivity 25mIU(hCG)/ml) is mandatory prior to inclusion and every month during the trial
14. Women of childbearing potential not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment. Male patients with a fertile partner are also required to secure effective methods of contraception (definition available in protocol)
15. Previous immunotherapy
16. Patients referred from a hospital outside of Denmark
17. Major dilation of veins or bowel obstructing the needle path
18. Persistent atrial fibrillation
19. Metal objects (e.g. biliary SEMS) within 5 cm of ablation target
20. Cardiac pacemaker or ICD, that cannot be safely disconnected during IRE treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | 6 months after treatment start
  (in patients receiving at least one dose of pembrolizumab, IRE and an evaluable CT-scan)
Serious adverse reaction (SAR) rate according to CTCAE v5 | cumulative after 12 months after treatment start
  (in patients receiving at least one dose of pembrolizumab)

SECONDARY OUTCOMES:
Median overall survival | Through study completion, an average of 1 year
Median progression-free survival | Through study completion, an average of 1 year
ORR | 2 months, 4 months and 6 months after treatment start
  (in patients that have received at least one dose of pembrolizumab and an evaluable CT-scan)
Clinical benefit ratio | 8 weeks after treatment start
  (defined as objective response or stable disease for at least 8 weeks during treatment in patients receiving at least one dose of pembrolizumab, IRE and an evaluable CT-scan)
Serum CA-19-9 response | 2 months, 4 months and 6 months after treatment start
  (response defined as a decrease of at least 20 % observed during treatment in patients with elevated CA 19-9 at baseline)
Survival rate | 6 months and 12 months after treatment start
Progression-free survival rate | 6 months and 12 months after treatment start
Mean difference in perceived quality of life measured by EORTC QLQ-C30 v3 | 2 months, 4 months, 6 months, 8 months, 10 months and 12 months after treatment start
  (for subscales: Global health status, Physical functioning, Fatigue, Nausea and vomiting, Pain, Appetite loss and Diarrhea)
Mean difference in nutrition status measured by PG-SGA-SF | 2 months, 4 months, 6 months, 8 months, 10 months and 12 months after treatment start
  (difference in total numerical score of the patient-generated subjective global assessment (short form) PG-SGA(c) SF (range 0-37, lower is better)
Difference in peripheral blood naïve T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood effector memory T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood central memory T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood effector T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood terminally differentiated effector T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood exhausted T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood regulatory T cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood conventional dendritic cell type 1 count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood conventional dendritic cell type 2 count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood plasmacytoid dendritic cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Difference in peripheral blood myeloid-derived suppressor cell count prior to IRE-treatment, 1 day after IRE-treatment and 6 weeks after IRE-treatment compared to baseline | 8 days, 11 days, 52 days after treatment start
  (based on flow cytometry measures of naïve, EM, CM, EFF, TE, EX T cells, Tregs, cDC1, cDC2, pDC and MDSC concentrations)
Histological tumor regression grade in tumor biopsies after pembrolizumab and after pembrolizumab + IRE compared to baseline | 10 days and 52 days after treatment start
  (based on the CAP regression grading system)
Difference in tumor RNA expression after pembrolizumab and after pembrolizumab + IRE compared to baseline | 10 days and 52 days after treatment start
  (based on NanoString RNA panCancer IO 360 gene panel. Analysis will explore the cancer-immunological mechanisms of the therapy in order to guide future studies. No specific outcomes are predetermined)
Difference in (histological) tumor infiltrating leukocyte (TIL) pattern after pembrolizumab and after pembrolizumab + IRE compared to baseline | 10 days and 52 days after treatment start
  (Based on analysis by immunohistochemistry. The relative concentration of leukocytes will be estimated and compared. The exact subpopulations of leukocytes will be based on the findings in outcomes 12 and 14, to validate the results)
Adverse event rate (CTCAEv5, all grades) | cumulative after 12 months after treatment start
  (all events registered during active treatment and follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ladekarl, DMSc, Principal Investigator — Department of Oncology
Locations (1):
- Department of Oncology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No